CLINICAL TRIAL: NCT01528904
Title: Fetal Thyroid Hormones Concentration In Hyperthyroid or Hypothyroid Pregnant Women
Brief Title: Maternal Autoimmune Thyroid Disease and Fetal Thyroxin
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Svetlana Spremovic Radjenovic, assistant professor, gynecologist and obstetrician, subspecialist in endocrinology, University of Belgrade
Other Study IDs: 318/VII-4/3 3186
Record Dates: First submitted 2012-01-12; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Pregnancy Complicated by Hyperthyroidism; Hypothyroidism in Pregnancy
Keywords: pregnancy; autoimmune thyroid disease; fetal thyroid hormones; antithyroid antibodies; ultrasound parameters

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hyperthyroid pregnant women: hyperthyroidism diagnosed and treated by an endocrinologist, based on clinical and laboratory tests and ultrasound thyroid examination.
- Hypothyroid pregnant women: hypothyroidism diagnosed and treated by an endocrinologist, based on clinical and laboratory tests and ultrasound thyroid examination
- Healthy pregnant women: uncomplicated pregnancies in healthy women, older then 35 years, directed for cordocentesis due to age, because of missed karyotyping in previous period of pregnancy

SUMMARY:
The purpose of this trial is to correlate fetal thyroid hormones from fetal cord blood with clinical (maternal antithyroid drug dose and antithyroid antibodies) and ultrasound (US) parameters of fetal thyroid function from pregnant mothers with autoimmune thyroid disease (AITD).

DETAILED DESCRIPTION:
Maternal hyperthyroidism in pregnancy is complicated with hypertension, preeclampsia, heart failure, thyroid storm, preterm labor and stillbirth, while the fetus suffers from intrauterine growth retardation (IUGR), goiter; neonatal prematurity and low birth weight.

Maternal hypothyroidism is seen in 2 % of pregnancies. Risks are higher for preeclampsia, postpartum hemorrhage, miscarriage, stillbirth, preterm birth and lower IQ score.

Thyroid stimulating hormone (TSH) receptor antibodies, antithyroid drugs and iodine pass to the fetus. So the fetus may also become a patient. Monitoring fetal growth, fetal heart rate (tachycardia is a late sign of fetal hyperthyroidism), bone maturation and the size of the fetal thyroid by ultrasound are important parameters for the assessment of transfer of hyperthyroidism from mother to the fetus

Patients follow up:

After inclusion into the study, thyroid function tests (fT4, TSH), and auto-antibodies assessment (anti TPO, TRAK) were performed once every two months in mothers with AITD, and from the 24th week of gestation monthly. Treatment was adjusted accordingly. Ultrasound for fetal size, morphology and fetal heart rate (FHR) was performed once in two months, and from the 24th week of gestation, monthly. The fetal biophysical profile score was determined weekly from the 30th week of gestation. The single centre design was chosen: all fetal sonograms were performed by the same gynecologist. Cardiotocography was performed once weekly from the 30th week of gestation.

Study design:

Fetal and maternal free thyroxin (fT4) and TSH, thyroid antibodies in mothers and fetal ultrasound (fetal size, morphology and fetal heart rate) were determined at the same time, once, from 22nd to 33rd weeks of gestation.

Procedure: Cordocentesis (Cordocentesis is a highly specialized prenatal test in which a fetal blood sample is removed from the umbilical cord and tested for genetic problems, hormones or infections. Cordocentesis can be done at 18 weeks of pregnancy or later). Fetal fT4 and TSH were measured from cord blood samples. Healthy pregnant subjects were directed for cordocentesis for karyotype analysis due to age (missed previous procedures for karyotyping).

The diagnosis of fetal hypo or hyperthyroidism was established taking into account fT4 concentrations according to the nomograms Thorpee-Beeston et al., 1996, 1991.

When fetal hyperthyroidism is diagnosed, antithyroid drugs given to the mother are administered or adjusted. When fetal hypothyroidism is diagnosed, then the possibility of intraamniotic thyroxin application is discussed with the mother.

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune hyper or hypothyroidism, diagnosed by an endocrinologist, treated, based on clinical and laboratory tests and ultrasound thyroid examination.
* Patients were included if they were seen by gynecologist at Clinic for Gynecology up until 20th week of gestation and not later.
* 20 healthy pregnant women in control group were directed for cordocentesis due to age.

Exclusion Criteria:

* Any other chronic diseases.

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Groups are selected from State tertiary referral centre for Gynecology and Obstetrics
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2001-01; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Fetal free thyroxin | 24th to 32nd week of gestation

SECONDARY OUTCOMES:
fetal ultrasound parameters | 24th to 32nd week of gestation
  at the same time as fetal free thyroxin sampling
maternal antithyroid antibodies | 24th to 32nd week of gestation
  sampled at the same time as the fetal free thyroxin
dose of maternal antithyroid medication (ATD) | 24th to 32nd week of gestation
  recorded at the same time as the fetal sampling for free thyroxin

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Spremovic-Radjenovic, MD PhD, Principal Investigator — Medical School of the University of Belgrade
Locations (1):
- Clinic for Gynecology and Obstetrics, Belgrade, Serbia, Serbia

REFERENCES:
- [Background] Abalovich M, Amino N, Barbour LA, Cobin RH, De Groot LJ, Glinoer D, Mandel SJ, Stagnaro-Green A. Management of thyroid dysfunction during pregnancy and postpartum: an Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2007 Aug;92(8 Suppl):S1-47. doi: 10.1210/jc.2007-0141. PMID 17948378